# **Clinical Trial Protocol:**

**Protocol Title:** A Randomized, Double-masked, Vehicle-controlled Study

Evaluating the Efficacy and Safety of Two Doses of OCS-01 compared to Vehicle in the Treatment of Inflammation and Pain Following Cataract Surgery

IND#

**Protocol Number:** DX216

Study Phase: 2

**Product Name:** OCS-01 ophthalmic suspension

**Indication:** Inflammation and pain following cataract surgery

**Investigator:** Multi-center clinical investigation

**Sponsor:** Oculis ehf.

Álfheimar 74, 6. hæð 104 Reykjavik | Iceland Tel. +354 546 4440

Contract Research

**Organizations:** 300 Brickstone Square

Andover, MA 01810

U.S.A

Ora, Inc.

Phone: +1-978-685-8900

| | Date |
|--------------------|----------------|
| Original Protocol: | 24 May 2019 |
| Amendment 1: | 08 August 2019 |

## **Confidentiality Statement**

This protocol contains confidential, proprietary information of Ora, Inc. and Oculis. Further dissemination, distribution, or copying of this protocol or its contents is strictly prohibited.


# **ORA PERSONNEL**

| <b>Department Sr. Vice President:</b> | _ |
|---------------------------------------|---|
| Project Manager: | |
| Medical Monitor | |


## 1 SYNOPSIS

Protocol Title: A Randomized, Double-masked, Vehicle-controlled Study

Evaluating the Efficacy and Safety of Two Doses of OCS-01 compared to Vehicle in the Treatment of Inflammation and Pain

Following Cataract Surgery

IND#

Protocol Number: DX216

Study Drugs: 1. OCS-01 (Dexamethasone Cyclodextrin Nanoparticle

Ophthalmic Suspension 1.5%)

2. Placebo (vehicle for OCS-01)

Study Phase: 2

**Objective(s):** The primary objective of this study is to evaluate the efficacy and

safety of OCS-01 once a day (QD) and twice a day (BID) compared to placebo (vehicle) BID in the treatment of inflammation and pain

following cataract surgery.

The secondary objective of this study is to evaluate the optimal dosing frequency of OCS-01 (QD versus BID) in the treatment of

inflammation and pain following cataract surgery.

Overall Study Design:

Structure: Multi-center, randomized, double-masked, placebo (vehicle)-

controlled study

**Duration:** Approximately 20-52 days

**Controls:** Placebo (vehicle for OCS-01)

groups

Dosage/Dose Regimen/

Instillation/

Application/Use:

Subjects will be randomized to one of the following treatment

Each subject will receive a master kit




# Summary of Visit Schedule:

Visit 1 (Day -28 to Day -1 [prior to surgery]): Screening, baseline evaluations

Visit 2 (Day 1 [18 to 30 hours post-surgery]): Review of inclusion and exclusion criteria, randomization, and dosing and dispensation of study medication

Visit 3 (Day 2) Pain assessments (telephone call)

Visit 4 (Day  $4\pm1$ ): Inflammation, pain, and safety assessments Visit 5 (Day  $8\pm1$ ): Inflammation, pain, and safety assessments Visit 6 (Day  $15\pm2$ ): Inflammation, pain, and safety assessments Visit 7 (Day  $22\pm2$ ): Inflammation, pain, and safety assessments, and exit visit

# Measures Taken to Reduce Bias:

Randomization will be used to avoid bias in the assignment of subjects to treatment, to increase the likelihood that known and unknown subject attributes (e.g. demographics and baseline characteristics) are evenly balanced across treatment groups, and to enhance the validity of statistical comparisons across treatment groups. Double-masked treatment will be used to reduce the potential of bias during data collection and the evaluation of clinical endpoints.

## **Study Population Characteristics:**

**Number of Subjects:** Approximately, 150 subjects will be randomized into the following groups:


Condition/ Disease:

Inflammation and pain following cataract surgery

**Inclusion Criteria:** 

Each subject must:

- 1. Provide written informed consent, approved by the appropriate ethics committee;
- 2. Be able to comply with the study requirements and visit schedule:
- 3. Be at least 18 years of age of either sex or any race;
- 4. Be planning to undergo unilateral cataract extraction via phacoemulsification and posterior chamber intraocular lens (PCIOL) implantation in the study eye;
- 5. Have an anterior chamber cell score
- 6. Have a pin-hole visual acuity (VA) without any other correction
- 7. Have a negative urine pregnancy test at Visit 1 (Day -1 to Day -28 [prior to surgery]), if female of childbearing potential (i.e. those who have experienced menarche, who are not surgically sterilized [bilateral tubal ligation, hysterectomy, or bilateral oophorectomy] or post-menopausal [12 months after last menses]) and must use acceptable effective contraceptive measure throughout the study period. Acceptable effective contraceptive measure is defined as hormonal oral, implantable, injectable, or transdermal contraceptives; mechanical spermicide in conjunction with a barrier such as condom or diaphragm; intrauterine device (IUD); or surgical sterilization of partner. For non-sexually active females, abstinence may be regarded as an adequate method of birth control.

## **Exclusion Criteria:**

## Each subject must not:

- Have a known sensitivity or allergy to dexamethasone, corticosteroids, or any of the study medication's components;
- 2. Be monocular;
- 3. Have any intraocular inflammation (e.g. white blood cells or flare) present in either eye at the Visit 1 (Day -1 to Day -28 [prior to surgery]) slit lamp examination;
- 4. Have a score on the Ocular Pain Assessment at Visit 1


- 5. Use anti-inflammatory agents, analgesics/pain relievers (including opioids, narcotics, and other pain medications), or immunomodulating agents, systemically or in either eye, and/or currently using or have any historic use of medications for benign prostatic hyperplasia (BPH)\_from the washout period through the duration of the study. Washout periods for medications prior to the day of cataract surgery are as follows:
  - a. Topical ocular steroids: 14 days;
  - b. Periocular injection of any corticosteroid solution: 28 days;
  - c. Intraocular treatment with a corticosteroid including dexamethasone drug delivery systems: 56 days after implantation; fluocinolone acetonide drug delivery systems: 48 months after implantation; any other intravitreal injection: 95 days after injection;

Note: While it is expected that subjects requiring an intraocular treatment with a corticosteroid will be excluded due to underlying exclusionary conditions, subjects who otherwise meet all eligibility criteria will be required to follow the above-mentioned washout intervals.

d. Any systemic treatment with a corticosteroid including oral: 14 days; systemic or parenteral sustained/extended release: 180 days;

Note: Inhaled, intranasal, and topical dermatologic steroids (except on the face and periocular region) are allowed. Topical dermatologic steroids on the face and periocular region require a 7 day washout.

- e. Topical ocular non-steroidal anti-inflammatory drugs (NSAIDs): 7 days;
- f. Systemic analgesics/pain relievers (e.g. gabapentin, pregabalin, and opioids): 14 days;

Note: Use of an opioid during cataract surgery is allowed;

g. Systemic acetaminophen, NSAIDs, acetylsalicylic acid, or other anti-inflammatory agents: 7 days;

Note: Use of up to 81 mg of acetylsalicylic acid dosed once daily is allowed if dosage has been stable for at least 30 days prior to surgery and will remain stable for the duration of the study.

- h. Medications for BPH (e.g. alpha adrenergic blocking agents including tamsulosin, silodosin, alfuzosin, and finasteride): all current or previous use of BPH medications excludes participation in this study.;
- i. Cyclosporine: 56 days or immunomodulating or immunosuppressive agents (e.g. calcineurin inhibitors, antiproliferative agents, mammalian target


- of rapamycin (mTOR) inhibitors, etc.): 2 months
- j. Mast cell stabilizers or antihistamines (e.g. β2adrenergic agonists. cromoglicic acid, ketotifen, brompheniramine, cetirizine, diphenhydramine): 7 days;
- 6. Require the use of a contact lens or a collagen shield within 72 hours prior to Visit 2 (Day 1 [18 to 30 hours post-surgery]) or for the remainder of the study period in either eye;
- 7. Require the use of non-diagnostic topical ophthalmic medications in either eye for the duration of the study with the exception of the following, which are allowed: mydriatics, anesthetics, antiseptics, balanced salt solution, viscoelastics, prophylactic antibiotics, non-prostaglandin analog intraocular pressure (IOP)-lowering agents, lid scrubs for mild blepharitis, or artificial tears for the management of dry eye (allowed topical medication should not be instilled at the same time as the study drug. Study medication should be instilled at least 30 minutes after any prior allowed topical medication. In addition, any other allowed topical medication should not be instilled within 2 hours following instillation of study medication);

#### 8. Have an IOP

surgery]).

Subjects taking IOP-lowering medication must not be on more than 1 IOP-lowering medication. Prostaglandin analogs are not allowed within 4 weeks of Visit 2 (Day 1 [18 to 30 hours post-

Note: Combination IOP agents count as 2 medications.

- 9. Currently have or have a history of herpes keratitis in the study eye;
- Have corneal abrasions or ulcers in the study eye (not including the surgical clear corneal wound from cataract surgery);
- 11. Have evidence of acute external ocular infections (bacterial, viral, and/or fungal such as vaccinia, varicella, and other viral diseases of the comea and conjunctiva), corneal endothelial dystrophies, intraocular infections, dysthyroid ophthalmopathy, active chalazion, or uncontrolled blepharitis in the study eye;
- 12. Have uncontrolled and clinically significant dry eye syndrome in the study eye (use of artificial tears is allowed);
- 13. Have active or a history of chronic or recurrent inflammatory eye disease (e.g. iritis, scleritis, uveitis, iridocyclitis, or rubeosis iritis) in either the fellow eye or the study eye;


- 14. Have cystoid macular edema, diabetic retinopathy, or diabetic macular edema; compromised macular function; significant macular diseases; or a history of macular edema in the study eye;
- 15. Have previous ocular trauma with visible scarring or any deformities due to the trauma in the study eye that in the opinion of the Investigator may affect the pharmacokinetics of the study medication, intraocular inflammation, or the normal healing process;
- 16. Have the potential for ocular hemorrhage in the study eye that may interfere with evaluation of post-surgery inflammation;
- 17. Have a planned use of femtosecond laser or any other ophthalmic surgical procedure (e.g. MIGS [minimally invasive glaucoma surgery], vitrectomy, relaxing incisions, iridectomy, conjunctival excisions, use of iris hooks or other iris dilators, etc.) in addition to the cataract extraction procedure via phacoemulsification and PCIOL implantation in the study eye;
- 18. Have a planned use of anterior capsule staining for capsulorhexis (i.e. trypan blue) during cataract surgery;
- 19. Have had corneal or retinal surgery (laser or incisional) in the study eye within 6 months of Visit 1 (Day -1 to Day -28 [prior to surgery]), or be planning to have laser or incisional surgery during the study period in the study eye (other than cataract surgery);
- 20. Have surgery planned or scheduled for the contralateral eye during the 3-week study period;
- 21. Have an immunosuppressive or an autoimmune disease that in the opinion of the Investigator could affect intraocular inflammation or the normal healing process of the eye;
- 22. Have active or chronic/recurrent ocular or systemic disease that is uncontrolled and will likely affect wound healing;
- 23. Currently have a suspected or known malignancy or be currently receiving anti-neoplastic therapy;
- 24. Have previously been enrolled in this clinical study, have planned to participate in another clinical trial during the follow-up period that could confound the treatment or outcomes of this investigation, or be currently in the follow-up period of a previous clinical trial;
- 25. Be enrolled in the study if the Investigator determines that the subject should not be included for reasons not already specified (e.g. systemic or other ocular disease/abnormality), if the health of the subject or the validity of the study outcomes may be compromised by the subject's enrollment;
- 26. Be a female who is currently pregnant, planning a


pregnancy, lactating, not using a medically acceptable form of birth control throughout the study duration, or have a positive urine pregnancy test at Visit 1 (Day -1 to Day -28 [prior to surgery]).

## **Evaluation Criteria:**

Hierarchical Primary Efficacy Measures:

**Efficacy Measures:** 

- 1. Absence of anterior chamber cells
- 2. Absence of pain

Secondary Efficacy Measures:

- Absence of anterior chamber cells at
- Absence of pain at
- Absence of flare at
- Absence of both anterior chamber cells and flare at
- Use of rescue medication on or prior to each visit and overall.
- Safety Measures:
- Change from baseline of pin-hole VA (without any other correction) as measured on the ETDRS chart;
- Change from baseline of IOP;
- Adverse event (AE) rates.
- **Rescue Criteria:**
- Grade anterior chamber cells
- Severe ocular pain at Visit 4 (Day 4) (or after) with oral acetaminophen.

## General Statistical Methods and Types of Analyses:




# Hypotheses

Primary Endpoint:



Hierarchical Primary Endpoint:



Sample Size Determination










# 2 TABLE OF CONTENTS

| 1 | SYN | OPSIS | 3 |
|---|------------|----------------------------------------------------|----|
| 2 | | LE OF CONTENTS | |
| | List | of Abbreviations | 16 |
| 3 | INTE | RODUCTION | 17 |
| | 3.1 | Background | 17 |
| | <b>3.2</b> | Study Rationale | 18 |
| | 3.3 | Dosage | 18 |
| | 3.4 | Placebo Justification | 19 |
| | 3.4.1 | Rationale | 19 |
| | 3.4.2 | Measures To Ensure Safe Participation in the Study | 20 |
| 4 | STU | DY OBJECTIVES AND HYPOTHESIS | 21 |
| | 4.1 | Study Objective | |
| | 4.2 | Study Hypothesis | |
| 5 | OVE | RALL STUDY DESIGN | 21 |
| 6 | STU | DY POPULATION | |
| | <b>6.1</b> | Number of Subjects (approximate) | |
| | <b>6.2</b> | Study Population Characteristics | |
| | 6.3 | Inclusion Criteria | |
| | <b>6.4</b> | Exclusion Criteria | |
| | 6.5 | Rescue Criteria | |
| | 6.6 | Withdrawal Criteria (if applicable) | |
| 7 | | DY PARAMETERS | |
| | <b>7.1</b> | Efficacy Measures | |
| | | 7.1.1 Primary Efficacy Measure | |
| | | 7.1.2 Secondary Efficacy Measure | |
| | | 7.1.3 Primary Efficacy Analyses | |
| | | 7.1.4 Secondary Efficacy Analyses | |
| | 7.2 | Safety Measures | |
| 8 | | DY MATERIALS | |
| | 8.1 | Study Treatment(s) | |
| | | 8.1.1 Study treatment(s) | |
| _ | | 8.1.2 Instructions for Use and Administration | |
| 9 | | DY METHODS AND PROCEDURES | |
| | 9.1 | Subject Entry Procedures | |
| | | 9.1.1 Overview | |
| | | 9.1.2 Informed Consent | |
| | | 9.1.3 Washout Intervals | |
| | | 9.1.4 Procedures for Final Study Entry | |
| | 0.2 | 9.1.5 Methods for Assignment to Treatment Groups: | |
| | 9.2 | Concurrent Therapies | |
| | | 9.2.1 Prohibited Medications/Treatments | |
| | | 9.2.2 Rescue Medications | |
| | | 9 / A Special Lifet of Activities | 30 |

| 9.3 | Examination Procedures | 30 |
|---|---|---|
| 9.4 | Schedule of Visits, Measurements and Dosing | |
| | 9.4.1 Scheduled Visits | |
| | 9.4.2 Unscheduled Visits | 33 |
| 9.5 | Compliance with Protocol | 33 |
| 9.6 | Subject Disposition | |
| | 9.6.1 Completed Subjects | 33 |
| | 9.6.2 Discontinued subjects | 33 |
| <b>9.7</b> | Study Termination | 34 |
| 9.8 | Study Duration | 34 |
| 9.9 | Monitoring and Quality Assurance | 34 |
| <b>ADV</b> | ERSE EVENTS | 34 |
| 10.1 | Adverse Event | 34 |
| | 10.1.1 Severity | 35 |
| | 10.1.2 Relationship to Study Drug | 35 |
| | 10.1.3 Expectedness | |
| 10.2 | Serious Adverse Events | |
| 10.3 | Procedures for Reporting Adverse Events | |
| | 10.3.1 Reporting a Suspected Unexpected Adverse Reaction | 37 |
| | 10.3.2 Reporting a Serious Adverse Event | |
| 10.4 | Procedures for Unmasking of Study Drug | 37 |
| 10.5 | Type and Duration of the Follow-up of Subjects after Adverse E | |
| STA' | TISTICAL METHODS | 38 |
| 11.1 | Statistical Hypotheses | |
| 11.2 | Analysis Populations | |
| 11.3 | Sample Size Determination | |
| 11.4 | Interim Analysis | |
| 11.5 | Efficacy Analysis | |
| | 11.5.1 General Statistical Considerations | |
| | 11.5.2 Primary Efficacy Analysis | 40 |
| | 11.5.3 Secondary Efficacy Analyses | 40 |
| 11.6 | Safety Analysis | |
| 11.7 | | |
| 11.8 | Demographics and Medical History | |
| | IPLIANCE WITH GOOD CLINICAL PRACTICES, ETHICAL | |
| | SIDERATIONS, AND ADMINISTRATIVE ISSUES | |
| | Protection of Human Subjects | |
| | 1 Subject Informed Consent | |
| | 12.1.2 Institutional Review Board Approval | |
| | 12.1.3 Ethical Conduct of the Study | |
| 12.2 | Subject Confidentiality | |
| | 12.3.1 Retention of Documentation. | |
| 12.4 | Labeling, Packaging, Storage, Accountability, and Return or Dis | |
| 1217 | Drug | _ |
| | 12.4.1 Labeling/Packaging | |
| | 12.7.1 Davening I dending | |

| | 12.4.2 Storage of Study Drug | 44 |
|------|-------------------------------------------------------------|----|
| | 12.4.3 Accountability of Study Drug | 44 |
| | 12.4.4 Return or Disposal of Study Drug | |
| 12.5 | Recording of Data on Source Documents and Case Report Forms | |
| | Handling of Biological Specimens | |
| | Publications | |
| | NCES | |
| | 1: Schedule of Visits and Measurements | |
| * * | 2: Examination Procedures, Tests, Equipment, and Techniques | |
| | 3: Protocol Amendment Summary | |
| | 4: Ora Approvals | |
| | 5: Investigator's Signature | |

#### List of Abbreviations

 $\gamma$ CD  $\gamma$ -cyclodextrin AE adverse event twice a day

BPH benign prostatic hyperplasia

CI confidence interval CD cyclodextrin

CFR Code of Federal Regulations eCRF electronic case report form EMA European Medicines Agency

ETDRS Early Treatment of Diabetic Retinopathy Study

FAS full analysis set

FDA Food and Drug Administration

GCP Good Clinical Practice
IB Investigator's Brochure
ICF informed consent form

ICH International Conference on Harmonisation

IOP intraocular pressure IRB institutional review board

IUD intrauterine device

LOCF last observation carried forward
MIGS minimally invasive glaucoma surgery
mTOR mammalian target of rapamycin
NSAID non-steroidal anti-inflammatory drug
PCIOL Posterior chamber intraocular lens

PI Principal Investigator

PP per protocol
PT preferred term
QD once a day

SAE serious adverse event SAP statistical analysis plan SOC system organ class

TEAE treatment-emergent adverse events

VA visual acuity


## 3 INTRODUCTION

## 3.1 Background

An estimated 95 million people worldwide are affected by cataracts, with cataract surgery being the most commonly performed surgical procedure in many countries (Liu, Wilkins et al. 2017). The current preferred treatments for ocular inflammation include the use of topical corticosteroids and/or non-steroidal anti-inflammatory drugs (NSAIDs), which may be contraindicated in some populations. Corticosteroids, which are considered the mainstay treatment for ocular inflammation, can be associated with adverse events (AEs), especially when frequent or prolonged dosing is needed, such as in patients where post-operative inflammation is severe and/or prolonged (Weber, Kodjikian et al. 2013).

In general, drug penetration from the ocular surface via topical administration into the eye encounters multiple barriers. This results in a bioavailability inside the eye that is generally well below 5%. In spite of this very low topical bioavailability, aqueous eye drops are the patient-preferred dosage form, especially in treatment of diseases of the anterior eye tissues, accounting for over 90% of the market (Loftsson and Stefansson 2017).

Dexamethasone is a corticosteroid that has been used in the form of eye drops (Maxidex®, Alcon, United States of America) to treat inflammation caused by surgery, infections, or injury (Alcon Laboratories 2002). Dexamethasone has limited solubility in water and does not readily permeate from the eye's aqueous exterior into the eye. Studies have shown that cyclodextrins (CDs) are able to enhance topical bioavailability of dexamethasone from aqueous eye drops (Usayapant, Karara et al. 1991, Kristinsson, Fridriksdottir et al. 1996, Sigurdsson, Konraethsdottir et al. 2007, Loftsson and Stefansson 2017). CDs have also been incorporated into other Food and Drug Administration (FDA) approved ophthalmic drops to increase drug solubility (Alcon Laboratories 2000). Oculis is developing a novel drug delivery platform composed of the active ingredient, dexamethasone, and CD nanoparticles (OCS-01, previously called DexNP), which aid in delivery of the active pharmaceutical ingredient from the ocular surface to both the anterior and posterior segments of the eye. CD-based dexamethasone eye drop solutions have been tested in human patients and show excellent penetration into the anterior segment of the eye (Kristinsson, Fridriksdottir et al. 1996, Saari, Nelimarkka et al. 2006, Tanito, Hara et al. 2011). Some of the earliest formulations of dexamethasone CD solutions (0.32) or 0.67% dexamethasone, 2-hydroxypropyl-β-cyclodextrin), were tested in a clinical trial conducted in Iceland 20 years ago (Kristinsson, Fridriksdottir et al. 1996). In 125 patients undergoing cataract surgery, concentrations of dexamethasone were significantly higher after application of dexamethasone CD suspension compared to Maxidex® (P < 0.001), indicating that the CD-based drug delivery system enhances both the solubility and permeability of dexamethasone to the anterior segment of the human eye. Notably, no toxic effects were observed with the use of dexamethasone CD suspension.

In a more recent study (Johannesson, Moya-Ortega et al. 2014), levels of dexamethasone were assessed in the tear fluid of healthy subjects treated with a topical application of 1.5% DexNP or Maxidex®. Six (6) subjects received DexNP in one eye and Maxidex® in the contralateral eye. Results reveal that treatment with DexNP results in a 19-fold higher concentration of dexamethasone compared to treatment with Maxidex®. Notably, 4 hours post-instillation, the


concentration of dexamethasone from DexNP treatment was still 10-times higher than what was observed with Maxidex® treatment. These results demonstrate that dexamethasone, complexed with CD nanoparticles, elicits a higher concentration and longer duration of action in the tear fluid than the currently available product, Maxidex®. Importantly, DexNP was well tolerated by the subjects and no serious adverse events (SAEs) were observed.

A study conducted by Saari et al. (Saari, Nelimarkka et al. 2006) evaluated the efficacy of an eye drop containing 0.7% dexamethasone-CD suspension, applied once daily, compared to a 0.1% dexamethasone sodium phosphate eye drops, applied three times daily for the treatment of post-operative inflammation after cataract surgery. The dexamethasone-CD suspension was shown to be safe and more effective in treating post-operative inflammation, after once daily dosing, than 0.1% dexamethasone sodium phosphate eye drops applied three times daily.

In the human studies with DexNP to date, DexNP was well tolerated and the only AE reported has been a modest rise in intraocular pressure (IOP), a known side effect of dexamethasone use, which subsided following discontinuation of DexNP in all cases (Kristinsson, Fridriksdottir et al. 1996) (Johannesson, Moya-Ortega et al. 2014) (Saari, Nelimarkka et al. 2006) (Tanito, Hara et al. 2011) (Ohira, Hara et al. 2015) (Krag and Hessellund 2014) (Shulman, Johannesson et al. 2015).

Building on the enhanced ocular penetration of DexNP, as well as its favorable efficacy results and safety profile, Oculis has developed an updated formulation, OCS-01, consisting of water soluble 1.5% Dexamethasone-yCD complexes to treat post-surgical inflammation.

## 3.2 Study Rationale

The trial outlined here is a randomized, double-masked, placebo (vehicle)-controlled study evaluating the efficacy and safety of two doses of OCS-01 compared to vehicle in the treatment of inflammation and pain following cataract surgery. The primary objective is to evaluate the efficacy and safety of OCS-01 compared to placebo and the secondary objective is to evaluate the optimal dosing frequency (once a day [QD] or twice a day [BID]).

#### 3.3 Dosage



As a comparison, Maxidex 0.1% dexamethasone suspension is an FDA approved ophthalmic suspension for the treatment of steroid responsive inflammatory conditions of the palpebral and bulbar conjunctiva, cornea, and anterior segment of the globe, including inflammation post-cataract surgery. In severe disease, 1-2 drops may be dosed hourly. A 0.1% suspension would contain 0.03 mg of dexamethasone per drop. If the maximum daily dose is applied, this would equate to 2 drops per hour, up to 48 drops. This could result in a maximum daily dose of 1.44 mg.


Further, the of dexamethasone per drop for OCS-01 is also assuming that the entire drop is absorbed into the eye. The maximum capacity of the conjunctival sac is up to and a drop of larger volume applied to a human eye will have its excess overflowed. Thus, a maximum of dexamethasone per drop will reach the eye.

The dexamethasone formulation to be tested here contains natural  $\gamma$ -cyclodextrin ( $\gamma$ CD).  $\gamma$ CD has been evaluated previously in other dexamethasone based eye drops (DexNP) in several indications in clinical trials (Tanito, Hara et al. 2011, Johannesson, Hallberg et al. 2014, Ohira, Hara et al. 2015, Shulman, Johannesson et al. 2015). The eye drops were well tolerated and displayed no signs of irritation or redness.

#### 3.4 Placebo Justification

This justification is based on Oculis' interpretation and position with regard to the International Conference on Harmonisation (ICH) Topic E10 guideline on the "Choice of control group in clinical trials" (CPMP/ICH/364/96).

## 3.4.1 Rationale

The inclusion of a placebo group is considered essential to the design of the DX216 study as:

- It provides the most rigorous evaluation of the efficacy and safety of OCS-01.
- It is required by the FDA as a negative control in post-cataract inflammation studies.
- It will allow indirect comparisons with Loteprednol and other studies that were recently conducted with a placebo design (Rajpal, Fong et al. 2013, Fong, Silverstein et al. 2018).

The sponsor believes that placebo can be safely and ethically administered in this study with close monitoring and rescue criteria based on the following rationale:

Guideline 5 of the International Ethical Guidelines for Health-related Research Involving Humans specifies that a placebo-controlled trial is acceptable only if "delaying or withholding the established effective intervention will result in no more than a minor increase above minimal risk to the participant and risks are minimized, including through the use of effective mitigation procedures" (CIOMS 2016). For this indication, pain and inflammation following cataract surgery, delaying or withholding intervention will not pose substantial risk to the subject. Further, there are rescue criteria defined in the protocol if the subject is displaying Grade 2 or greater anterior cells or experiencing severe ocular pain.

Protocol Section 6.5: Rescue Criteria:




In addition, several studies have been completed in both Europe and in the US to evaluate a study drug for ocular pain and inflammation using a placebo-controlled trial design. Some examples include:

**NCT00198445:** Safety and Efficacy Study of Topical Bromfenac Versus Placebo to Treat Ocular Inflammation After Cataract Surgery

**NCT01367249:** Efficacy of Bromfenac Ophthalmic Solution in Patients Undergoing Cataract Surgery

NCT01426854: Nepafenac Compared to Placebo for Ocular Pain and Inflammation

NCT01318499: Nepafenac 0.3% Two Study

**NCT00405730:** Nepafenac 0.1% Eye Drops, Suspension Compared to Ketorolac Trometamol 0.5% Eye Drops, Solution and Placebo

**NCT00430092:** Difluprednate 0.5% Eye Drops Compared to Placebo for Inflammation Following Ocular Surgery

**NCT02208297:** Lotemax 0.38% Gel Compared to Placebo for Inflammation and Pain Following Cataract Surgery

## 3.4.2 Measures To Ensure Safe Participation in the Study

Placebo-controlled studies may only be ethically conducted when patients at a controlled risk are included, patients are fully informed of all the potential risks, patients are carefully monitored, and adequate protocol safety measures are in place. In this proposed trial a number of general protective measures are incorporated into the study protocol with the intention to minimize the risk to patients.

The following specific measures are included in the protocol:

- Patients at low risk are selected and they will be fully informed of their chances of randomization to the placebo group during informed consent.
- Patients are carefully monitored for pain and inflammation following cataract surgery.
- The rescue and withdrawal criteria minimize patients risk and will allow proper medical care.

Based on the above rationale and the measurements for a safe medical supervision for the patients, Oculis believes that it is scientifically and ethically appropriate to use placebo control in the study DX216.


## 4 STUDY OBJECTIVES AND HYPOTHESIS

## 4.1 Study Objective

The primary objective of this study is to evaluate the efficacy and safety of OCS-01 QD and BID compared to placebo (vehicle) BID in the treatment of inflammation and pain following cataract surgery.

The secondary objective of this study is to evaluate the optimal dosing frequency of OCS-01 (QD versus BID) in the treatment of inflammation and pain following cataract surgery.

## 4.2 Study Hypothesis

It is hypothesized that

## 5 OVERALL STUDY DESIGN

This is a multi-center, randomized, double-masked, placebo (vehicle)-controlled study, designed to evaluate the efficacy and safety of OCS-01 ophthalmic suspension (QD versus BID) compared to placebo in treating inflammation and pain following cataract surgery.



#### 6 STUDY POPULATION

## 6.1 Number of Subjects (approximate)

Approximately 150 subjects will be enrolled in the study.

This is a multi-center study.

# 6.2 Study Population Characteristics

Subjects may be of either sex or any race and must be at least 18 years of age at Visit 1 (Day -1 to Day -28 [prior to surgery]). Subjects must be planning to undergo unilateral cataract extraction via phacoemulsification and posterior chamber intraocular lens (PCIOL) implantation in the study eye and must meet all of the inclusion criteria and none of the exclusion criteria.


#### 6.3 Inclusion Criteria

## Each subject must:

- 1. Provide written informed consent, approved by the appropriate ethics committee;
- 2. Be able to comply with the study requirements and visit schedule;
- 3. Be at least 18 years of age of either sex or any race;
- 4. Be planning to undergo unilateral cataract extraction via phacoemulsification and PCIOL implantation in the study eye;
- 5. Have an anterior chamber cell score6. Have a pin-hole visual acuity (VA) without any other correction
- 7. Have a negative urine pregnancy test at Visit 1 (Day -1 to Day -28 [prior to surgery]), if female of childbearing potential (i.e. those who have experienced menarche, who are not surgically sterilized [bilateral tubal ligation, hysterectomy, or bilateral oophorectomy] or post-menopausal [12 months after last menses]) and must use acceptable effective contraceptive measure throughout the study period. Acceptable effective contraceptive measure is defined as hormonal oral, implantable, injectable, or transdermal contraceptives; mechanical spermicide in conjunction with a barrier such as condom or diaphragm; intrauterine device (IUD); or surgical sterilization of partner. For non-sexually active females, abstinence may be regarded as an adequate method of birth control.

#### 6.4 Exclusion Criteria

## Each subject must <u>not</u>:

- 1. Have a known sensitivity or allergy to dexamethasone, corticosteroids, or any of the study medication's components;
- 2. Be monocular;
- 3. Have any intraocular inflammation (e.g. white blood cells or flare) present in either eye
- 4. Have a score on the Ocular Pain Assessment at


- 5. Use anti-inflammatory agents, analgesics/pain relievers (including opioids, narcotics, and other pain medications), or immunomodulating agents, systemically or in either eye, and/or currently using or have any history of use of medications for benign prostatic hyperplasia (BPH) from the washout period through the duration of the study. Washout periods for medications prior to the day of cataract surgery are as follows:
  - a. Topical ocular steroids: 14 days;
  - b. Periocular injection of any corticosteroid solution: 28 days;
  - c. Intraocular treatment with a corticosteroid including dexamethasone drug delivery systems: 56 days after implantation; fluocinolone acetonide drug delivery systems: 48 months after implantation; any other intravitreal injection: 95 days after injection;

Note: While it is expected that subjects requiring an intraocular treatment with a corticosteroid will be excluded due to underlying exclusionary conditions, subjects who otherwise meet all eligibility criteria will be required to follow the above-mentioned washout intervals.

d. Any systemic treatment with a corticosteroid including oral: 14 days; systemic or parenteral sustained/extended release: 180 days;

Note: Inhaled, intranasal, and topical dermatologic steroids (except on the face and periocular region) are allowed. Topical dermatologic steroids on the face and periocular region require a 7 day washout.

- e. Topical ocular NSAIDs: 7 days;
- f. Systemic analgesics/pain relievers (e.g. gabapentin, pregabalin, and opioids): 14 days;

Note: Use of an opioid during cataract surgery is allowed;

g. Systemic acetaminophen, NSAIDs, acetylsalicylic acid, or other antiinflammatory agents: 7 days;

Note: Use of up to 81 mg of acetylsalicylic acid dosed once daily is allowed if dosage has been stable for at least 30 days prior to surgery and will remain stable for the duration of the study.

- h. Medications for BPH (e.g. alpha adrenergic blocking agents including tamsulosin, silodosin, alfuzosin, and finasteride): all current or previous use of BPH medications excludes participation in this study.;
- i. Cyclosporine: 56 days or immunomodulating or immunosuppressive agents (e.g. calcineurin inhibitors, antiproliferative agents, mammalian target of rapamycin (mTOR) inhibitors, etc.): 2 months
- j. Mast cell stabilizers or anti-histamines (e.g. β2-adrenergic agonists. cromoglicic acid, ketotifen, brompheniramine, cetirizine, diphenhydramine): 7 days;
- 6. Require the use of a contact lens or a collagen shield within 72 hours prior to Visit 2 (Day 1 [18 to 30 hours post-surgery]) or for the remainder of the study period in either eye;


- 7. Require use of non-diagnostic topical ophthalmic medications in either eye for the duration of the study with the exception of the following, which are allowed: mydriatics, anesthetics, antiseptics, balanced salt solution, viscoelastics, prophylactic antibiotics, non-prostaglandin analog IOP-lowering agents, lid scrubs for mild blepharitis, or artificial tears for the management of dry eye (allowed topical medication should not be instilled at the same time as the study drug. Study medication should be instilled at least 30 minutes after any prior allowed topical medication. In addition, any other allowed topical medication should not be instilled within 2 hours following instillation of study medication);
- 8. Have an IOP
  Subjects taking IOP-lowering medication must not be on more than 1 IOP-lowering medication. Prostaglandin analogs are not allowed within 4 weeks of Visit 2 (Day 1 [18 to 30 hours post-surgery]).

Note: Combination IOP agents count as 2 medications.

- 9. Currently have or have a history of herpes keratitis in the study eye;
- 10. Have corneal abrasions or ulcers in the study eye (not including the surgical clear corneal wound from cataract surgery);
- 11. Have evidence of acute external ocular infections (bacterial, viral, and/or fungal such as vaccinia, varicella, and other viral diseases of the cornea and conjunctiva), corneal endothelial dystrophies, intraocular infections, dysthyroid ophthalmopathy, active chalazion, or uncontrolled blepharitis in the study eye;
- 12. Have uncontrolled and clinically significant dry eye syndrome in the study eye (use of artificial tears is allowed);
- 13. Have active or a history of chronic or recurrent inflammatory eye disease (e.g. iritis, scleritis, uveitis, iridocyclitis, or rubeosis iritis) in either the fellow eye or the study eye;
- 14. Have cystoid macular edema, diabetic retinopathy, or diabetic macular edema; compromised macular function; significant macular diseases; or a history of macular edema in the study eye;
- 15. Have previous ocular trauma with visible scarring or any deformities due to the trauma in the study eye that in the opinion of the Investigator may affect the pharmacokinetics of the study medication, intraocular inflammation, or the normal healing process;
- 16. Have the potential for ocular hemorrhage in the study eye that may interfere with evaluation of post-surgery inflammation;
- 17. Have a planned use of femtosecond laser or any other ophthalmic surgical procedure (e.g. minimally invasive glaucoma surgery [MIGS], vitrectomy, relaxing incisions, iridectomy, conjunctival excisions, use of iris hooks or other iris dilators, etc.) in addition to the cataract extraction procedure via phacoemulsification and PCIOL implantation in the study eye;
- 18. Have a planned use of anterior capsule staining for capsulorhexis (i.e. trypan blue) during cataract surgery;


- 19. Have had corneal or retinal surgery (laser or incisional) in the study eye within 6 months of Visit 1 (Day -1 to Day -28 [prior to surgery]), or be planning to have laser or incisional surgery during the study period in the study eye (other than cataract surgery);
- 20. Have surgery planned or scheduled for the contralateral eye during the 3-week study period;
- 21. Have an immunosuppressive or an autoimmune disease that in the opinion of the Investigator could affect intraocular inflammation or the normal healing process of the eye;
- 22. Have active or chronic/recurrent ocular or systemic disease that is uncontrolled and will likely affect wound healing;
- 23. Currently have a suspected or known malignancy or be currently receiving anti-neoplastic therapy;
- 24. Have previously been enrolled in this clinical study, have planned to participate in another clinical trial during the follow-up period that could confound the treatment or outcomes of this investigation, or be currently in the follow-up period of a previous clinical trial:
- 25. Be enrolled in the study if the Investigator determines that the subject should not be included for reasons not already specified (e.g. systemic or other ocular disease/abnormality), if the health of the subject or the validity of the study outcomes may be compromised by the subject's enrollment;
- 26. Be a female who is currently pregnant, planning a pregnancy, lactating, not using a medically acceptable form of birth control throughout the study duration, or have a positive urine pregnancy test at Visit 1 (Day -1 to Day -28 [prior to surgery]).

## 6.5 Rescue Criteria

- Grade anterior chamber cells

  [see Appendix 2: Examination Procedures, Tests, Equipment, and Techniques])
- Severe ocular pain

  Examination Procedures, Tests, Equipment, and Techniques])

## 6.6 Withdrawal Criteria (if applicable)

Any subject who wishes to withdraw from the study for any reason is entitled to do so at any time without obligation.

Any subject who discontinues study drug or who is administered rescue therapy will remain enrolled in the study and continue to participate in all subsequent visits for safety and efficacy assessments. If a subject discontinues participation in the study early, every attempt will be made to complete the exit procedures required at the final study visit (Visit 7).


is

#### 7 STUDY PARAMETERS

## 7.1 Efficacy Measures

#### 7.1.1 Primary Efficacy Measure

Hierarchical Primary Efficacy Measures:

- 1. Absence of anterior chamber cells
- 2. Absence of pain

## 7.1.2 Secondary Efficacy Measure

Secondary Efficacy Measures:

- Absence of anterior chamber cells
- Absence of pain
- Absence of flare
- Absence of <u>both</u> anterior chamber cells and flare
- Use of rescue medication on or prior to each visit and overall.

#### 7.1.3 Primary Efficacy Analyses

The hierarchical primary efficacy analyses are as follows:

1. Difference between the two treatment arms in the proportion of study eyes with absence of anterior chamber cells

If the proportion of study eyes with absence of anterior chamber cells statistically significantly higher for OCS-01 versus placebo (vehicle)

2. Difference in the proportion of study eyes with absence of pain

#### 7.1.4 Secondary Efficacy Analyses

- <u>Difference in the proportion of study eyes with absence of anterior chamber cells</u>
- Difference in the proportion of study eyes with absence of pain
- Difference in the proportion of study eyes with absence of flare


- Difference in the proportion of study eyes with absence of both anterior chamber cells and anterior chamber flare
- Use of rescue medication on or prior to each visit and overall.

Efficacy measures will be further described in the Statistical Analysis Plan (SAP).

## 7.2 Safety Measures

Safety will be assessed by the following measures:

- Change from baseline of pin-hole VA (without any other correction) as measured on the ETDRS chart
- Change from baseline of IOP
- AE rates

## 8 STUDY MATERIALS

## 8.1 Study Treatment(s)

- 8.1.1 Study treatment(s)
  - OCS-01 ophthalmic suspension (QD) + Placebo (vehicle) (QD)
  - OCS-01 ophthalmic suspension (BID)
  - Placebo (vehicle) ophthalmic suspension (BID)
- 8.1.2 <u>Instructions for Use and Administration</u>

The master kit's

contents will be as follows for subjects randomized to each of the respective treatment arms:

- OCS-01 QD + Placebo (vehicle) QD
- OCS-01 BID
- Placebo (vehicle) BID


For all other study visits, subjects should continue to dose according to their established schedule. If the visit is scheduled during the time of normal dosing, the subject should bring their dose with them to the visit for administration. Every effort should be made to maintain dosing schedule/ frequency.

## 9 STUDY METHODS AND PROCEDURES

## 9.1 Subject Entry Procedures

## 9.1.1 Overview

Subjects as defined by the criteria in Sections 6.2, 6.3, and 6.4 will be considered for entry into this study.

#### 9.1.2 Informed Consent

Prior to a subject's participation in the trial (i.e. changes in a subject's medical treatment and/or study related procedures), the study will be discussed with each subject, and subjects wishing to participate must give informed consent (and/or assent) using an informed consent form (ICF). The ICF must be the most recent version that has received approval/favorable review by a properly constituted institutional review board (IRB).

#### 9.1.3 Washout Intervals

Washout periods are outlined in exclusion criteria in Section0.

#### 9.1.4 Procedures for Final Study Entry

Subjects must satisfy all of the inclusion and none of the exclusion criteria in order to be entered into the study.

#### 9.1.5 Methods for Assignment to Treatment Groups:

Each subject who signs an ICF will be assigned a screening number. Screening numbers will be assigned in sequential order at each site beginning with 001 and will follow the two-digit site number (e.g. subject 077 at Site 99 will have Screening Number 99-077). Inclusion and exclusion criteria will be reviewed, and qualifying subjects will be enrolled into the study. Each subject who qualifies for entry will be assigned a randomization number and corresponding treatment according to the randomization code. Study drug will be randomly assigned using , stratified by site, via an interactive response system.


## 9.2 Concurrent Therapies

The use of any concurrent medication, prescription, or over-the-counter, is to be recorded on the subject's source document and corresponding electronic case report form (eCRF) along with the reason the medication was taken.

Concurrent enrollment in another study drug or device study is not permitted.

#### 9.2.1 Prohibited Medications/Treatments

Prohibited medications and washout periods are summarized in Table 1.

- Ocular surgical intervention scheduled on the contralateral eye within 3 weeks post-cataract surgery; or corneal or retinal surgery (laser or incisional) in the study eye within 6 months of Visit 1 (Day -1 to Day -28 [prior to surgery]); or laser or incisional surgery during the study period in the study eye (other than cataract surgery);
- Use of a contact lens or a collagen shield 72 hours prior to Visit 2 (Day 1 [18 to 30 hours post-surgery]) and for the remainder of the study period in either eye;
- Use anti-inflammatory agents, analgesics/pain relievers (including opioids, narcotics, and other pain medications), or immunomodulating agents, systemically or in either eye, and/or currently using or have any historic use of medications for benign prostatic hyperplasia (BPH) from the washout period through the duration of the study;
- Non-diagnostic topical ophthalmic medications in either eye for the duration of the study with the exception of the following mydriatics, anesthetics, antiseptics, balanced salt solution, viscoelastics, prophylactic antibiotics, non-prostaglandin analog IOP lowering agents, lid scrubs, or artificial tears (allowed topical medication should not be instilled at the same time as the study drug. Study medication should be instilled at least 30 minutes after any prior allowed topical medication. In addition, any other allowed topical medication should not be instilled within 2 hours following instillation of study medication);
- Planned use of anterior capsule staining for capsulorhexis (i.e. trypan blue) during cataract surgery;
- Concurrent enrollment or enrollment within the follow-up period in another study drug or device study is not allowed.

**Table 1: Non-allowed Medications and Washout Periods** 

| Medication | Washout Period |
|---|---|
| Topical ocular steroids | 14 days |
| Periocular injection of any corticosteroid solution | 28 days |
| Intraocular treatment with a corticosteroid | 56 days after implantation |
| Fluocinolone acetonide drug delivery systems | 48 months after implantation |
| Intravitreal injection | 95 days after injection |
| Systemic treatment with a corticosteroid including oral | 14 days |
| Systemic or parenteral sustained/extended release corticosteroid | 180 days |
| Topical ocular NSAIDs | 7 days |
| Systemic analgesics/pain relievers (e.g. gabapentin, pregabalin, and opioids) | 14 days |


| Systemic acetaminophen, NSAIDs, acetylsalicylic acid, or other anti-inflammatory | 7 days |
|---|---|
| agents | |
| BPH medication (e.g. alpha adrenergic blocking agents including tamsulosin, silodosin, alfuzosin, and finasteride) | _no current or historic use |
| Immunomodulating or immunosuppressive agents (e.g. cyclosporine, calcineurin inhibitors, antiproliferative agents, mTOR inhibitors, etc.) | 56 days |
| Mast cell stabilizers or anti-histamines (e.g. β2-adrenergic agonists. cromoglicic acid, ketotifen, brompheniramine, cetirizine, diphenhydramine) | 7 days |

#### 9.2.2 Rescue Medications



• Severe ocular pain [see Appendix 2: Examination Procedures, Tests, Equipment, and Techniques])

## 9.2.3 Special Diet or Activities

There are no special diet or activity restrictions for this study.

#### 9.3 Examination Procedures

Procedures to be performed at each study visit with regard to the study objectives are detailed in Appendix 2: Examination Procedures, Tests, Equipment, and Techniques.

## Visit 1 — Screening and Baseline Evaluations (-28 to -1 days prior to surgery)

- Informed consent/assent
- Demographic data
- Medical and medication history
  - Current underlying conditions, including those that began within the last 30 days, which may have been resolved before Visit 1 (Day -1 to Day -28 [prior to surgery]), must be recorded.
  - Any medications the subject is taking, as well as those the subject may have taken but discontinued within 30 days prior to Visit 1 (Day -1 to Day -28 [prior to surgery]) must be recorded.
- Urine pregnancy test (if applicable)
- Inclusion/exclusion criteria
- Ocular pain (study eye only)
- Pin-hole VA
- Slit lamp biomicroscopy


- Ocular inflammation assessment of the anterior chamber cell and flare (study eye only)
- IOP
- Dilated indirect ophthalmoscopy

## Visit 2 — Day 1 (18 to 30 hours post-surgery)

- Review inclusion/exclusion criteria
- Medical and medications update
- Ocular pain (study eye only)
- Pin-hole VA
- Slit lamp biomicroscopy
- Ocular inflammation assessment of the anterior chamber cell and flare (study eye only)
- Randomization
- Dose and dispense study medication and dosing diary
- Query for AEs

## Visit 3 — Day 2 (Telephone Call)

• Ocular pain (study eye only)

## Visit 4 — Day 4 (± 1 day window)

- Medical and medications update
- Ocular pain (study eye only)
- Pin-hole VA
- Slit Lamp Biomicroscopy
- Ocular inflammation assessment of the anterior chamber cell and flare (study eye only)
- IOP
- Query for AE

## Visit 5 — Day 8 ( $\pm$ 1 day window)

- Medical and medications update
- Ocular pain (study eye only)
- Pin-hole VA
- Slit lamp biomicroscopy
- Ocular inflammation assessment of the anterior chamber cell and flare (study eye only)


- IOP
- Query for AEs

## Visit 6 — Day 15 ( $\pm$ 2 day window)

- Medical and medications update
- Ocular pain (study eye only)
- Pin-hole VA
- Slit lamp biomicroscopy
- Ocular inflammation assessment of the anterior chamber cell and flare (study eye only)
- IOP
- Query for AEs

## Visit 7 — Day 22 ( $\pm$ 2 day window)

- Urine pregnancy test (if applicable)
- Medical and medications update
- Ocular pain (study eye only)
- Pin-hole VA
- Slit lamp biomicroscopy
- Ocular inflammation assessment of the anterior chamber cell and flare (study eye only)
- IOP
- Dilated indirect ophthalmoscopy
- Query for AEs
- Exit from study

AEs (both elicited and observed) will be monitored throughout the study. All AEs (both elicited and observed) will be promptly reviewed by the Investigator for accuracy and completeness. All AEs will be documented on the appropriate eCRF.

If a female has a positive pregnancy test during the study, then the Investigator will notify the site's monitor immediately. The Investigator shall request from the subject and/or the subject's physician copies of all related medical reports during the pregnancy and shall document the outcome of the pregnancy. The Investigator will retain these reports together with the subject's source documents and will provide a copy of all documentation to the site's monitor.


## 9.4 Schedule of Visits, Measurements and Dosing

#### 9.4.1 Scheduled Visits

Refer to Appendix 1: Schedule of Visits and Measurements for a schedule of visits and measurements

## 9.4.2 Unscheduled Visits

In the case of an AE, an unscheduled visit may occur. The Investigator may perform additional assessments at their discretion. All additional assessments will be documented in the subject's source document and eCRF.

## 9.5 Compliance with Protocol

This study will be conducted in compliance with the protocol, the ethical principles that have their origin in the Declaration of Helsinki, and the ICH consolidated Guideline E6 for Good Clinical Practice (GCP) (European Medicines Agency/ Committee for Medicinal Products for Human Use/ICH/135/1995).

## 9.6 Subject Disposition

## 9.6.1 Completed Subjects

A completed subject is defined as having completed all 7 visits. Subjects who have discontinued from the study or withdrawn consent/assent will not be considered completed subjects.

#### 9.6.2 Discontinued subjects

Subjects may be discontinued prior to their completion of the study due to the following:

- AEs
- Protocol violations
- Subject's decision (e.g. withdrawal of consent)
- Administrative reasons (e.g. inability to continue, lost to follow up)
- Sponsor termination of study
- Principal Investigator's (PI) decision
- other

Note: In addition, any subject may be discontinued for any sound medical reason.

If at any time during the study the Investigator deems that the subject's safety has been compromised or the subject has been non-compliant, the subject may be withdrawn from the study.


Any subject who wishes to withdraw from the study for any reason is entitled to do so at any time without obligation.

Notification of a subject's discontinuation and the reason for discontinuation will be made to Ora and/or the Sponsor and will be clearly documented on the eCRF.

Any subject who discontinues study drug or who is administered rescue therapy will remain enrolled in the study and continue to participate in all subsequent visits for safety and efficacy assessments. If a subject discontinues participation in the study early, every attempt will be made to complete the exit procedures required at the final study visit (Visit 7).

# 9.7 Study Termination

The study may be stopped at any time by the Investigator (at their respective site), the Sponsor, and/or Ora with appropriate notification.

# 9.8 Study Duration

Subjects may be screened from Day -28 to Day -1 prior to surgery. The study will involve 7 visits including a follow-up visit at Visit 7 (Day 22). Overall study duration will be 20-52 days, including the screening visit and a follow-up visit.

## 9.9 Monitoring and Quality Assurance

During the course of the study an Ora monitor, or designee, will make routine site visits to review protocol compliance, assess test article accountability, and ensure the study is being conducted according to the pertinent regulatory requirements. The review of the subjects' medical records will be performed in a manner to ensure that data protection and subject confidentiality rights are adequately maintained. Further details of the study monitoring will be outlined in a Monitoring Plan.

Regulatory authorities of domestic and foreign agencies, Ora Quality Assurance, and/or its designees may carry out on-site inspections and/or audits that may include source data checks. Therefore direct access to the original source data will be required for inspections and/or audits. All inspections and/or audits will be carried out giving consideration to data protection as well as subject confidentiality to the extent that local, national, and international laws apply.

#### 10 ADVERSE EVENTS

#### **10.1 Adverse Event**

An AE is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not the event is considered drug-related. An AE can therefore be any unfavorable and unintended sign (e.g. an abnormal laboratory finding), symptom, or disease occurring after the subject started dosing with the study drug, without any judgment about causality. Any pre-existing medical condition that worsens after administration of the study drug will also be considered a new AE. Study drug includes the study drug under evaluation (OCS-01)


and any comparator drug, placebo (vehicle), or any other medications required by the protocol given during any stage of the study.

Documentation regarding the AE should be made as to the nature, date of onset, end date, severity, relationship to study drug, action(s) taken, seriousness, and outcome of any sign or symptom observed by the physician or reported by the subject upon indirect questioning.

## <u>10.1.1</u> Severity

Severity of an AE is defined as a qualitative assessment of the degree of intensity of an AE as determined by the Investigator or reported to him/her by the subject. The assessment of severity is made irrespective of the relationship to study drug or the seriousness of the event and should be evaluated according to the following scale:

- *Mild:* AE is noticeable to the subject, but is easily tolerated and does not interfere with the subject's daily activities.
- *Moderate*: AE is bothersome, possibly requiring additional therapy, and may interfere with the subject's daily activities.
- Severe: AE is intolerable, necessitates additional therapy or alteration of therapy, and interferes with the subject's daily activities.

## 10.1.2 Relationship to Study Drug

The relationship of each AE to the study drug should be determined by the Investigator using these explanations:

- Suspected: A reasonable possibility exists that the study drug caused the AE.
- *Not Suspected:* A reasonable possibility does not exist that the study drug caused the AE.

"Suspected adverse reaction" means any AE for which there is a reasonable possibility that the study drug caused the AE. "Reasonable possibility" means there is evidence to suggest a causal relationship between the study drug and the AE. Types of evidence that would suggest a causal relationship between the study drug and the AE include: a single occurrence of an event that is uncommon and known to be strongly associated with drug exposure (e.g. angioedema, hepatic injury, Stevens-Johnson Syndrome); one or more occurrences of an event that is not commonly associated with drug exposure, but is otherwise uncommon in the population exposed to the drug (e.g. tendon rupture); an aggregate analysis of specific events observed in a clinical trial (such as known consequences of the underlying disease or condition under investigation or other events that commonly occur in the study population independent of drug therapy) that indicates those events occur more frequently in the drug treatment group than in a concurrent or historical control group.

#### 10.1.3 Expectedness

The expectedness of an AE should be determined based upon existing safety information about the study drug using these explanations:


- *Unexpected:* an AE that is not listed in the Investigator's Brochure (IB) or is not listed at the specificity or severity that has been observed.
- Expected: an AE that is listed in the IB at the specificity and severity that has been observed.

AEs that are mentioned in the IB as occurring with a class of drugs or as anticipated from the pharmacological properties of the drug, but are not specifically mentioned as occurring with the particular drug under investigation are to be considered unexpected.

Preliminary determination of classification of an AE as unexpected is the responsibility of the Investigator and subject to the Medical Monitor's final determination.

#### **10.2** Serious Adverse Events

An AE is considered serious if, in the view of either the Investigator or Sponsor, it results in any of the following outcomes:

- Death:
- A life-threatening AE;

Note: An AE is considered "life-threatening" if, in the view of either the Investigator or Sponsor, its occurrence places the subject at immediate risk of death. It does not include an AE that, had it occurred in a more severe form, might have caused death.

• Inpatient hospitalization or prolongation of existing hospitalization;

Note: The term "inpatient hospitalization" refers to any inpatient admission (even if less than 24 hours). For chronic or long-term inpatients, inpatient admission includes transfer within the hospital to an acute/intensive care inpatient unit. Inpatient hospitalization does not include: emergency room visits; outpatient/same-day/ambulatory procedures; observation/short stay units; rehabilitation facilities; hospice facilities; nursing homes; or clinical research/Phase 1 units.

Note: The term "prolongation of existing hospitalization" refers to any extension of an inpatient hospitalization beyond the stay anticipated or required for the reason for the initial admission as determined by the Investigator or treating physician.

• A persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions;

Note: A SAEs specifically related to visual threat would be interpreted as any potential impairment or damage to the subject's eyes (e.g., hemorrhage, retinal detachment, central corneal ulcer, or damage to the optic nerve).

• A congenital anomaly/birth defect.

Important medical events that may not result in death, are life-threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they


may jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.

#### **10.3 Procedures for Reporting Adverse Events**

All AEs and their outcomes must be reported to Ora, the study Sponsor, and the IRB as required by the IRB, federal, state, or local regulations and governing health authorities and recorded on the appropriate eCRF.

#### 10.3.1 Reporting a Suspected Unexpected Adverse Reaction

All AEs that are 'suspected' and 'unexpected' are to be reported to Ora, the study Sponsor, and the IRB as required by the IRB, regional and local regulations, and governing health authorities.

#### 10.3.2 Reporting a Serious Adverse Event

To ensure subject safety, all SAEs, regardless of their relationship to the study drug, must be immediately reported. All information relevant to the SAE must be recorded on the appropriate case report forms. The Investigator is obligated to pursue and obtain information requested by Ora and/or the Sponsor in addition to that information reported on the case report form. All subjects experiencing an SAE must be followed-up with and the outcome reported.

In the event of an SAE, the Investigator must notify Ora and the Sponsor upon becoming aware of a SAE; obtain and maintain in his/her files including all pertinent medical records, information, and medical judgments from colleagues who assisted in the treatment and follow-up of the subject; provide Ora and the study Sponsor with a complete case history, which includes a statement as to whether the event was or was not suspected to be related to the use of the study drug; and inform the IRB of the AE within their guidelines for reporting SAEs.

Investigators are to contact the study's Medical Monitor or designee upon becoming aware of a SAE.

#### 10.4 Procedures for Unmasking of Study Drug

The randomization code should be broken only in the event of a medical emergency, or when knowing the treatment assignment is absolutely necessary for the medical management of the study subject. When possible (i.e. in non-emergency situations), the study Sponsor or representative should be notified prior to unmasking study drug. In emergency situations, the Investigator must notify the Sponsor within 24 hours after determining that it is necessary to unmask the treatment assignment. The Investigator must also indicate in source documents and in the eCRF that the mask was broken and provide the date, time, and reason for breaking the mask. Any AE or SAE associated with breaking the mask must be recorded and reported as specified in this protocol.

#### 10.5 Type and Duration of the Follow-up of Subjects after Adverse Events

AEs will be followed until the condition is resolved or stabilized.


# 11 STATISTICAL METHODS

A complete detailed description of the statistical methods will be provided in the SAP.

# 11.1 Statistical Hypotheses

The hierarchical statistical hypotheses for evaluating the objectives of the study are as follows:

Primary Endpoint:



Hierarchical Primary Endpoint:






# 11.2 Analysis Populations

The following analysis populations will be defined, although additional populations and further refinement of the below populations may be specified in the SAP, prior to unmasking study data:



# 11.4 Interim Analysis

Interim analyses will not be performed.


# 11.5 Efficacy Analysis

#### 11.5.1 General Statistical Considerations



# 11.5.2 Primary Efficacy Analysis

**Primary Efficacy Measure:** The hierarchical primary efficacy measures are the absence of anterior chamber cells

**Primary Efficacy Analysis:** The primary efficacy variables, the absence of anterior chamber cells at Visit 6 (Day 15) and the absence of pain at Visit 4 (Day 4),

#### 11.5.3 Secondary Efficacy Analyses

Secondary Efficacy Measure: The secondary efficacy measures include:

1. Absence of anterior chamber cells

2. Absence of pain

3. Absence of flare


| 4. Absence of both anterior chamber cells and flare |
|---|
| 5. Use of rescue medication on or prior to each visit and overall. |
| Secondary Efficacy Analysis: The secondary efficacy variables, the differences in proportions of: study eyes with absence of anterior chamber cells study eyes with absence of pain study eyes with absence of both anterior chamber cells and anterior chamber flare will be summarized and analyzed similarly to the primary efficacy summaries and analyses. |
| Use of rescue medication on or prior to each visit will be |
| 11.6 Safety Analysis |
| The primary safety analyses will summarize VA, IOP, and AEs, as described below. |
| Appendix 2: Examination Procedures, Tests, Equipment, and Techniques. |
| Appendix 2: Examination Procedures, Tests, Equipment, and Techniques. |

# 11.7 Handling of Missing Data

The primary analyses of all efficacy data will use last observation carried forward (LOCF) to impute missing data; data for visits after a subject is discontinued for lack of efficacy or receives


rescue medication will be imputed as failures for success/failure endpoints and will be imputed using LOCF for other endpoints. To check robustness of results, sensitivity analyses of the primary efficacy endpoints will include analyses of observed data only, imputing data from subject visits after discontinuation for lack of efficacy or receipt of rescue medication as failures. Tipping point analysis and multiple imputation methods using monotone methodology will also be used to impute missing data as additional sensitivity analyses. PP analyses will use observed data only, with the exception of subjects who have missing data due to discontinuation for lack of efficacy or for subjects who receive rescue medication; for these subjects, missing data after discontinuation or data after receiving rescue medication will be imputed as failures for success/failure endpoints and will be imputed using LOCF for other endpoints.

#### 11.8 Demographics and Medical History

Subject demographics comprising age, gender, race, and ethnicity will be presented using discrete or continuous summary statistics as appropriate.

# 12 COMPLIANCE WITH GOOD CLINICAL PRACTICES, ETHICAL CONSIDERATIONS, AND ADMINISTRATIVE ISSUES

This study will be conducted in compliance with the protocol, with GCPs including ICH Guidelines, and in general, consistent with the Declaration of Helsinki. In addition, all applicable local, state, and federal requirements relevant to the use of study drugs in the countries involved will be adhered to.

#### 12.1 Protection of Human Subjects

#### 12.1.1 Subject Informed Consent

Informed consent must take place before any study specific procedures are initiated. Signed and dated written informed consent must be obtained from each subject prior to enrollment into the study.

All ICFs must be approved for use by the Sponsor and receive approval/favorable opinion from an IRB prior to their use. If the consent form requires revision (e.g., due to a protocol amendment or significant new safety information), it is the investigator's responsibility to ensure that the amended informed consent is reviewed and approved by Ora prior to submission to the governing IRB and that it is read, signed and dated by all subjects subsequently enrolled in the study as well as those currently enrolled in the study.

#### 12.1.2 <u>Institutional Review Board Approval</u>

This study is to be conducted in accordance with IRB regulations (U.S. 21 Code of Federal Regulations [CFR] Part 56.103). The Investigator must obtain appropriate IRB approval before initiating the study and re-approval at least annually.

Only an IRB approved version of the ICF will be used.


#### 12.1.3 Ethical Conduct of the Study

This study will be conducted in accordance with the ethical principles that originated with the Declaration of Helsinki.

#### 12.2 Subject Confidentiality

All personal study subject data collected and processed for the purposes of this study should be maintained by the Investigator and his/her staff with adequate precautions as to ensure that the confidentiality of the data in accordance with local, state, and federal laws and regulations.

Monitors, auditors and other authorized representatives of Ora, the Sponsor, the IRB approving this study, the FDA, the Department of Health and Human Services, other domestic government agencies, and other foreign regulatory agencies will be granted direct access to the study subject's original medical and study records for verification of the data and/or clinical trial procedures. Access to this information will be permitted to the aforementioned individuals to the extent permitted by law.

A report of the results of this study may be published or sent to the appropriate health authorities in any country in which the study drug may ultimately be marketed, but the subject's identity will not be disclosed in these documents.

#### 12.3 Documentation

Source documents may include a subject's medical records, hospital charts, clinic charts, the Investigator's study subject files, as well as the results of diagnostic tests such as X-rays, laboratory tests, and electrocardiograms. The Investigator's copy of the eCRF serves as the Investigator's record of a subject's study-related data.

#### 12.3.1 Retention of Documentation

All study related correspondence, subject records, consent forms, record of the distribution and use of all study drug and copies of case report forms should be maintained on file for at least two years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region; or until at least two years have elapsed since the formal discontinuation of clinical development of the study drug. These documents will be retained for a longer period if required by the applicable regulatory requirements or by an agreement with the Sponsor. It is the responsibility of the Sponsor to inform the investigator/institution as to when these documents no longer need to be retained.

If the responsible Investigator retires, relocates, or for other reasons withdraws from the responsibility of keeping study records, custody must be transferred to a person who will accept the responsibility. The Sponsor must be notified in writing of the name and address of the new custodian.


# 12.4 Labeling, Packaging, Storage, Accountability, and Return or Disposal of Study Drug

#### 12.4.1 Labeling/Packaging

All study drugs will be labeled according to applicable regulatory requirements.

#### 12.4.2 Storage of Study Drug

The study drug must be stored in a secure area accessible only to the Investigator and his/her designees. The study drug will be dispensed only to subjects entered into the clinical study, in accordance with the conditions specified in this protocol.

Once dispensed to subjects, study drug should be stored at ambient temperature.

#### 12.4.3 Accountability of Study Drug

The study drug is to only be prescribed by the PI or his/her named sub Investigator(s), and is to only be used in accordance with this protocol. The study drug must only be distributed to subjects eligible under this protocol to receive study drug.

The Investigator or his/her designee must keep an accurate accounting of the study drug received from the supplier. This includes the amount of study drug dispensed to subjects, amount of study drug returned to the Investigator by the subjects, and the amount returned or disposed upon the completion of the study. A detailed inventory must be completed for the study drug.

#### 12.4.4 Return or Disposal of Study Drug

At the end of the study, all study drugs will be returned to the Sponsor or their designee or destroyed at the study site. The return or disposal of study drug will be specified in writing.

#### 12.5 Recording of Data on Source Documents and Case Report Forms

All subject data will be captured in the subject source documents which will be transcribed in the eCRFs. The Investigator is responsible for ensuring that study data is completely and accurately recorded on each subject's eCRF, source documents, and all study-related materials. All study data should also be attributable, legible, contemporaneous, and original. Recorded datum should only be corrected in a manner that does not obliterate, destroy, or render illegible the previous entry (e.g., by drawing a single line through the incorrect entry and writing the revision next to the corrected data). An individual who has corrected a data entry should make clear who made the correction and when, by adding to the correction his/her initials as well as the date of the correction.

Data entry of all enrolled and randomized subjects will use software that conforms to 21 CFR Part 11 requirements, and will be performed only by staff who have been trained on the system


and have access to the system. Data will not be entered for screen failure subjects. An audit trail will be maintained within the electronic system to capture all changes made within the eCRF database. After the end of the study and database lock, compact discs (CDs) containing copies of all applicable subjects' eCRFs will be provided to each Investigator Site to be maintained on file by the Investigator.

# 12.6 Handling of Biological Specimens

Not applicable

#### 12.7 Publications

Authorship and manuscript composition will reflect joint cooperation among all parties involved in the study. Authorship will be established prior to the writing of the manuscript. The study Sponsor will have the final decision regarding the manuscript and publication.


#### REFERENCES

Alcon Laboratories, I. (2000). PAZEO (olopatadine hydrochloride ophthalmic solution) 0.7%.

Alcon Laboratories, I. (2002). Maxidex 0.1 % (dexamethasone ophthalmic suspension).

CIOMS (2016). International Ethical Guidelines for Health-related Research Involving Humans. Geneva.

Fong, R., B. E. Silverstein, J. H. Peace, J. I. Williams and J. L. Vittitow (2018). "Submicron loteprednol etabonate ophthalmic gel 0.38% for the treatment of inflammation and pain after cataract surgery." J Cataract Refract Surg 44(10): 1220-1229.

Jabs, D. A., R. B. Nussenblatt, J. T. Rosenbaum and G. Standardization of Uveitis Nomenclature Working (2005). "Standardization of uveitis nomenclature for reporting clinical data. Results of the First International Workshop." Am J Ophthalmol **140**(3): 509-516.

Johannesson, G., P. Hallberg, A. Eklund, A. Behndig and C. Linden (2014). "Effects of topical anaesthetics and repeated tonometry on intraocular pressure." <u>Acta Ophthalmol</u> **92**(2): 111-115.

Johannesson, G., M. D. Moya-Ortega, G. M. Asgrimsdottir, S. H. Lund, M. Thorsteinsdottir, T. Loftsson and E. Stefansson (2014). "Kinetics of gamma-cyclodextrin nanoparticle suspension eye drops in tear fluid." Acta Ophthalmol **92**(6): 550-556.

Krag, S. and A. Hessellund (2014). "Topical dexamethasone-cyclodextrin microparticle eye drops for uveitic macular oedema." <u>Acta Ophthalmol</u> **92**(8): e689-690.

Kristinsson, J. K., H. Fridriksdottir, S. Thorisdottir, A. M. Sigurdardottir, E. Stefansson and T. Loftsson (1996). "Dexamethasone-cyclodextrin-polymer co-complexes in aqueous eye drops. Aqueous humor pharmacokinetics in humans." <u>Invest Ophthalmol Vis Sci</u> **37**(6): 1199-1203.

Liu, Y. C., M. Wilkins, T. Kim, B. Malyugin and J. S. Mehta (2017). "Cataracts." <u>Lancet</u> **390**(10094): 600-612.

Loftsson, T. and E. Stefansson (2017). "Cyclodextrins and topical drug delivery to the anterior and posterior segments of the eye." <u>Int J Pharm</u> **531**(2): 413-423.

McCaffery, M. and A. Beebe (1994). "Pain: clinical manual for nursing practice." <u>Nurs Stand</u> **9**(11): 55.

Ohira, A., K. Hara, G. Johannesson, M. Tanito, G. M. Asgrimsdottir, S. H. Lund, T. Loftsson and E. Stefansson (2015). "Topical dexamethasone gamma-cyclodextrin nanoparticle eye drops increase visual acuity and decrease macular thickness in diabetic macular oedema." <u>Acta Ophthalmol</u> **93**(7): 610-615.


- Rajpal, R. K., R. Fong and T. L. Comstock (2013). "Loteprednol etabonate ophthalmic gel 0.5% following cataract surgery: integrated analysis of two clinical studies." <u>Adv Ther</u> **30**(10): 907-923
- Saari, K. M., L. Nelimarkka, V. Ahola, T. Loftsson and E. Stefansson (2006). "Comparison of topical 0.7% dexamethasone-cyclodextrin with 0.1% dexamethasone sodium phosphate for postcataract inflammation." <u>Graefes Arch Clin Exp Ophthalmol</u> **244**(5): 620-626.
- Samudre, S. S., F. A. Lattanzio, Jr., P. B. Williams and J. D. Sheppard, Jr. (2004). "Comparison of topical steroids for acute anterior uveitis." J Ocul Pharmacol Ther **20**(6): 533-547.
- Shulman, S., G. Johannesson, E. Stefansson, A. Loewenstein, A. Rosenblatt and Z. Habot-Wilner (2015). "Topical dexamethasone-cyclodextrin nanoparticle eye drops for non-infectious Uveitic macular oedema and vitritis a pilot study." Acta Ophthalmol **93**(5): 411-415.
- Sigurdsson, H. H., F. Konraethsdottir, T. Loftsson and E. Stefansson (2007). "Topical and systemic absorption in delivery of dexamethasone to the anterior and posterior segments of the eye." <u>Acta Ophthalmol Scand</u> **85**(6): 598-602.
- Tanito, M., K. Hara, Y. Takai, Y. Matsuoka, N. Nishimura, P. Jansook, T. Loftsson, E. Stefansson and A. Ohira (2011). "Topical dexamethasone-cyclodextrin microparticle eye drops for diabetic macular edema." <u>Invest Ophthalmol Vis Sci</u> **52**(11): 7944-7948.
- Usayapant, A., A. H. Karara and M. M. Narurkar (1991). "Effect of 2-hydroxypropyl-beta-cyclodextrin on the ocular absorption of dexamethasone and dexamethasone acetate." <u>Pharm Res</u> **8**(12): 1495-1499.
- Weber, M., L. Kodjikian, F. E. Kruse, Z. Zagorski and C. M. Allaire (2013). "Efficacy and safety of indomethacin 0.1% eye drops compared with ketorolac 0.5% eye drops in the management of ocular inflammation after cataract surgery." Acta Ophthalmol **91**(1): e15-21.


**Appendix 1: Schedule of Visits and Measurements** 



# Appendix 2: Examination Procedures, Tests, Equipment, and Techniques

| Pin-hole Visual Acuity | . 50 |
|---|---|
| Slit-lamp Evaluation | . 52 |
| During Slit Lamp Biomicroscopy: Ocular Inflammation Assessment of the Anterior Chamber | |
| Cell and Flare (Study Eye Only). | |
| Ocular Pain Grading Scale (Study Eye Only) | |
| Intraocular Pressure Procedures | |
| Dilated Indirect Ophthalmoscopy | 56 |


# Pin-hole Visual Acuity







# **Slit-lamp Evaluation**




# <u>During Slit Lamp Biomicroscopy: Ocular Inflammation Assessment of the Anterior Chamber Cell and Flare (Study Eye Only)</u>




# Ocular Pain Grading Scale (Study Eye Only)




# Intraocular Pressure Procedures




# **Dilated Indirect Ophthalmoscopy**




#### APPENDIX 3: PROTOCOL AMENDMENT SUMMARY

#### AMENDMENT 1

BACKGROUND AND RATIONALE FOR AMENDMENT



#### SUMMARY OF CHANGES

In the table below, the protocol text was amended by the following conventions:

- Deletions to the original text are indicated by strike through letters.
- Additions to amended text are indicated by bold letters.
- Replacements of wording in the amended text are indicated by bold and italicized letters.





# Appendix 4: Ora Approvals

**Protocol Title:** 

A Randomized, Double-masked, Vehicle-Controlled Study

Evaluating the Efficacy and Safety of Two Doses of OCS-01 compared to Vehicle in the Treatment Inflammation and Pain

Following Cataract Surgery

**Protocol Number:** 

DX216

**Protocol Date:** 

08Aug2019

This clinical study protocol was subject to critical review and has been approved by the Sponsor. The following personnel contributed to writing and/or approving this protocol.



### **Appendix 5: Investigator's Signature**

**Protocol Title:** A Randomized, Double-masked, Vehicle-Controlled Study Evaluating

the Efficacy and Safety of Two Doses of OCS-01 compared to Vehicle in the Treatment Inflammation and Pain Following Cataract Surgery

**Protocol Number:** DX216 **Protocol Date:** 08Aug2019

I agree to implement and conduct the study diligently and in strict compliance with the protocol, good clinical practices and all applicable laws and regulations. I agree to maintain all information supplied by the Sponsor and its agents in confidence and, when this information is submitted to an Institutional Review Board (IRB), Ethical Review Committee (ERC) or another group, it will be submitted with a designation that the material is confidential.

I have read this protocol in its entirety, including the above statement, and I agree to all aspects.

| Signed: | Date: |
|-------------------|-------|
| Name: | |
| Title: | |
| Affiliation: | |
| Address: | |
| Telephone number: | |

